CLINICAL TRIAL: NCT06401889
Title: Enhancing Skin Appearance and Quality of Life in Breast Cancer Survivors on Aromatase Inhibitor Therapy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC220302; NCI-2024-03468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-002971 (Other: Mayo Clinic Institutional Review Board); MC220302 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Adenocarcinoma; Estrogen Receptor-Positive Breast Carcinoma; Progesterone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete surveys/questionnaires, undergo skin measurement with the VISIA CA device, undergo facial skin photography, and attend consultations with an aesthetician on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates changes in skin quality and self-esteem among breast cancer patients who are initiating aromatase inhibitor therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the incidence and severity of skin quality changes after initiation of Aromatase Inhibitor (AI) therapy in breast cancer (BC) survivors through use of Canfield Sciences VISIA-CA technology and facial skin assessment photography.

II. Evaluate impact of AI therapy on patient-reported self-esteem and dermatology related life quality through validated patient reported outcome measures.

III. Assess for objective improvements in skin quality measurements with VISIA-CA after skincare intervention with aesthetician consultation.

IV. Measure changes in patient-reported self-esteem and dermatology related life quality following skincare intervention.

OUTLINE: This is an observational study.

Patients complete surveys/questionnaires, undergo skin measurement with the VISIA CA device, undergo facial skin photography, and attend consultations with an aesthetician on study.

ELIGIBILITY:
Inclusion Criteria:

* * Female ≥ 18 years

  * Postmenopausal women suitable to receive aromatase inhibitor as per physician's discretion
  * Histologically confirmed adenocarcinoma of the breast stage 0-III with estrogen receptor (ER) and/or progesterone receptor (PR) positive per American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) guideline and any human epidermal growth factor receptor 2 (HER2)
  * Patients must not have received any prior chemotherapy or endocrine therapy for their current breast cancer. Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer may be included
  * Patients willing to avoid any facial procedures including facials, neurotoxin injections, fillers, or lasers during study period
  * Willing and able to provide consent

Exclusion Criteria:

* * Patients who have previously taken AIs

  * Patients using prescription tretinoin, neurotoxin injections, fillers, facial lasers, microneedling, or facials within 6 months of study consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 years or older with diagnosis of estrogen receptor (ER) positive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in skin quality | Up to 6 months
  Changes in skin quality measured as incidence and severity of skin quality changes using VISIA-CA technology (skin analysis imaging system) and facial skin assessment photography.

CONTACTS AND LOCATIONS:
Overall Officials: Leila M. Tolaymat, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials